CLINICAL TRIAL: NCT07075289
Title: Comparing Oral Lumbrokinase DLBS1033 and Betahistine Mesylate in Benign Paroxysmal Positional Vertigo: A Randomized Comparative Study on Inflammatory Markers, Quality of Life, and Symptom Resolution
Brief Title: Comparing Oral Lumbrokinase DLBS1033 and Betahistine Mesylate in Benign Paroxysmal Positional Vertigo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitas Sebelas Maret (Other)
Collaborators: Dexa Medica Group (Industry)
Responsible Party: Principal Investigator, Stefanus Erdana Putra, Medical Doctor (Neurologist), Universitas Sebelas Maret
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 623/II/HREC/2024; UST-002.24/DLBS1033/1/2024 (Other Grant/Funding Number: Dexa Medica)
Record Dates: First submitted 2025-07-01; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Benign Paroxysmal Positional Vertigo (Disorder)
Keywords: benign paroxysmal positional vertigo (BPPV); betahistine mesylate; dizziness; inflammation; oral lumbrokinase DLBS1033; quality of life
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo; Dizziness; Inflammation | interventions — DLBS 1033; Betahistine

STUDY DESIGN:
Intervention Model Description: This study was designed as a randomized controlled double-masked trial, representing a robust experimental approach to compare the therapeutic effects of oral lumbrokinase DLBS1033 (490 mg, DISOLF film-coated tablet, Dexa Medica b.i.d.) and betahistine mesylate (12 mg, MERTIGO SR tablet, Dexa Medica b.i.d.) in patients suffering from BPPV for a 14-day prospective observation period. The research was carried out at the Neurology Outpatient Clinic of Dr. Moewardi General Hospital in Surakarta, Central Java, Indonesia, between April and August 2024, following full ethical approval from the hospital's Health Research Ethics Committee.
Who Masked: Participant, Investigator
Masking Description: The study protocol involved a two-block randomization to ensure balanced group assignments. The random sequences for the group allocation were generated by independent personnel of the direct study management and kept in sealed envelopes. This allocation concealment ensured that neither the investigator team nor the participants knew their assigned treatment. Each package was coded with the subject identification number according to the generated random number and assigned to each eligible subject. These codes remained unrevealed until the study's completion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral lumbrokinase DLBS1033 group (Experimental): BPPV patients who got oral lumbrokinase DLBS1033 (490 mg, DISOLF film-coated tablet, Dexa Medica b.i.d.) for 14-day prospective observation period.
  Interventions: Drug: DLBS1033
- Betahistine mesylate group (Active Comparator): BPPV patients who got betahistine mesylate (12 mg, MERTIGO SR tablet, Dexa Medica b.i.d.) for 14-day prospective observation period.
  Interventions: Drug: Betahistine Mesylate tablet

INTERVENTIONS:
Drug: DLBS1033 — Participants would get oral lumbrokinase DLBS1033 (490 mg, DISOLF film-coated tablet, Dexa Medica b.i.d.) for a 14-day prospective observation period.
  Arms: Oral lumbrokinase DLBS1033 group
Drug: Betahistine Mesylate tablet — Patients would get betahistine mesylate (12 mg, MERTIGO SR tablet, Dexa Medica b.i.d.) for a 14-day prospective observation period.
  Arms: Betahistine mesylate group

SUMMARY:
The goal of this clinical trial is to learn if oral lumbrokinase DLBS1033 works better than betahistine mesylate on inflammation, quality of life, and dizziness symptoms of adult benign paroxysmal positional vertigo (BPPV) patients. It will also learn about the safety of oral lumbrokinase DLBS1033 as a causative therapy of BPPV. The main questions it aims to answer are:

* Is there a difference in the decrease in IL-1β levels between BPPV patients who receive oral lumbrokinase DLBS1033 therapy and patients who receive betahistine mesylate therapy?
* Is there a difference in the decrease in TNF-α levels between BPPV patients who receive oral lumbrokinase DLBS1033 therapy and patients who receive betahistine mesylate therapy?
* Is there a difference in the decrease in VCAM-1 levels between BPPV patients who receive oral lumbrokinase DLBS1033 therapy and patients who receive betahistine mesylate therapy?
* Is there a difference in the quality of life between BPPV patients who receive oral lumbrokinase DLBS1033 therapy and patients who receive betahistine mesylate therapy?
* Is there a difference in the time to improve dizziness symptoms between BPPV patients who receive oral lumbrokinase DLBS1033 therapy and patients who receive betahistine mesylate therapy? Researchers will compare oral lumbrokinase DLBS1033 to betahistine mesylate to see if oral lumbrokinase DLBS1033 works better to treat BPPV

Participants will:

* Join a brief interview to find out the current and past medical history, as well as a physical examination of the study participants
* Give blood samples for biomarker examination, which will be conducted at the Clinical Pathology Laboratory of Dr. Moewardi Surakarta Hospital
* Take oral lumbrokinase DLBS1033 or betahistine mesylate every day for 2 weeks
* Visit the clinic once every week for evaluation and the blood test
* Keep a diary of their symptoms

DETAILED DESCRIPTION:
This study was designed as a randomized controlled double-masked trial, representing a robust experimental approach to compare the therapeutic effects of oral lumbrokinase DLBS1033 (490 mg, DISOLF film-coated tablet, Dexa Medica b.i.d.) and betahistine mesylate (12 mg, MERTIGO SR tablet, Dexa Medica b.i.d.) in patients suffering from BPPV for a 14-day prospective observation period. The research was carried out at the Neurology Outpatient Clinic of Dr. Moewardi General Hospital in Surakarta, Central Java, Indonesia, between April and August 2024, following full ethical approval from the hospital's Health Research Ethics Committee.

The study population comprised patients attending the aforementioned clinic, with specific inclusion and exclusion criteria applied to select eligible subjects via a purposive sampling method. Included patients were between 18 and 65 years old, diagnosed with BPPV by a neurologist based on a clear history of positional vertigo symptoms (nausea, vomiting, imbalance with head movements) and characteristic torsional nystagmus during the Dix-Hallpike maneuver (latency, fatigability, duration less than 60 seconds). Furthermore, participants had to be proficient in Indonesian and provide informed consent. Patients were excluded if they were pregnant or breastfeeding, showed signs of central vertigo or other neurological deficits, had current ear infections, hearing impairment, tinnitus, head trauma, or underlying conditions such as thyroid disorders, diabetes mellitus, osteoarthritis, a history of neoplasm, cardiovascular disease, hypertension, or recent ear/mastoid surgery. Cognitive impairment and participation in other clinical trials within 30 days prior to screening were also grounds for exclusion. To ensure data integrity, dropout criteria were established for patients unable to complete the study protocol, those who did not adhere to procedures, or those failing to complete the necessary questionnaires.

A total of 44 participants were enrolled, determined by a sample size calculation based on a 95% confidence interval and 5% confidence limits, with an additional 10% allowance for potential dropouts from a previous year's patient population of 751 peripheral vertigo cases. Standardized instruments were utilized for data collection, including the Indonesian version of Dizziness Handicap Inventory (DHI) for assessing quality of life which categorize it as poor, moderate, or good based on physical, emotional, and functional aspects; and the Indonesian version of the Vertigo Symptom Scale-Short Form (VSS-SF) to evaluate dizziness symptom severity, which is categorized as severe or low [15]. Furthermore, concentrations of key inflammatory biomarkers, specifically TNF-α, IL-1β, and VCAM-1, were quantified using Human Quantikine R&D Systems kits on a Thermo Fisher Invitrogen auto-analyzer according to manufacturer specifications.

The study protocol involved a two-block randomization to ensure balanced group assignments. The random sequences for the group allocation were generated by independent personnel of the direct study management and kept in sealed envelopes. This allocation concealment ensured that neither the investigator team nor the participants knew their assigned treatment. Each package was coded with the subject identification number according to the generated random number and assigned to each eligible subject. These codes remained unrevealed until the study's completion. The investigator team members, assigned as the enumerators, conducted symptom and quality of life assessments using the DHI and VSS-SF on the first day (baseline), seventh day, and fourteenth day after treatment initiation. Concurrently, blood samples were collected to assess TNF-α, IL-1β, and VCAM-1 levels. All collected data were then compiled and statistically analyzed using SPSS for Windows 25.0. Before hypothesis testing, data completeness and accuracy were verified, followed by coding, tabulation, and entry into the software. Normality of data distribution was assessed using the Kolmogorov-Smirnov test. Independent T-tests were performed for normally distributed data. Multiple linear regression analysis was conducted to investigate the relationship between inflammatory markers, quality of life, and potential confounding variables, and ordinal logistic regression analysis was conducted to determine the odds ratios (ORs) for inflammation levels and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years old
* Diagnosed with BPPV by a neurologist based on a clear history of positional vertigo symptoms (nausea, vomiting, imbalance with head movements) and characteristic torsional nystagmus during the Dix-Hallpike maneuver (latency, fatigability, duration less than 60 seconds)
* Proficient in Indonesian
* Provided informed consent

Exclusion Criteria:

* Pregnant or breastfeeding
* Showed signs of central vertigo or other neurological deficits
* Had current ear infections, hearing impairment, tinnitus, head trauma, or underlying conditions such as thyroid disorders, diabetes mellitus, osteoarthritis, a history of neoplasm, cardiovascular disease, hypertension, or recent ear/mastoid surgery.
* Cognitive impairment
* Participation in other clinical trials within 30 days prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-12-27 (Actual)

PRIMARY OUTCOMES:
Dizziness severity | baseline, day 7, and day 14
  The total value obtained from filling in the Indonesian version of the Vertigo Symtom Scale-Short Version (VSS-SF) in BPPV patients which can reflect the severity of dizziness symptoms (floating, swinging or shifting sensations) in patients.
Quality of life from the BPPV patients | baseline, day 7, and day 14
  The total value obtained from filling in the Dizziness Handicap Inventory (DHI) questionnaire in BPPV patients which can reflect the impact of dizziness on the physical, emotional and functional aspects of the patient's daily life.
Inflammatory biomarkers of the BPPV patients | baseline, day 7, and day 14
  TNF-α, IL-1β, and VCAM-1 levels as pro-inflammatory biomarkers were measured before patients received therapy, on the 7th day after receiving therapy, and on the 14th day after patients received therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Stefanus E Putra, MD, Principal Investigator — Department of Neurology, Faculty of Medicine, Universitas Sebelas Maret
Locations (1):
- Dr. Moewardi Regional General Hospital, Surakarta, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Publication in ICMJE journals
Supporting Information: Study Protocol, SAP, CSR
Time Frame: July 1st, 2025-July 1st, 2026
Access Criteria: Open access, every journal visitor

REFERENCES:
- [Background] Walther LE, Wenzel A, Buder J, Bloching MB, Kniep R, Blodow A. Detection of human utricular otoconia degeneration in vital specimen and implications for benign paroxysmal positional vertigo. Eur Arch Otorhinolaryngol. 2014 Dec;271(12):3133-8. doi: 10.1007/s00405-013-2784-6. Epub 2013 Oct 30. PMID 24170182
- [Background] Tang Y, Zhou X, Cao T, Chen E, Li Y, Lei W, Hu Y, He B, Liu S. Endoplasmic Reticulum Stress and Oxidative Stress in Inflammatory Diseases. DNA Cell Biol. 2022 Nov;41(11):924-934. doi: 10.1089/dna.2022.0353. Epub 2022 Sep 14. PMID 36356165
- [Background] Bashiruddin J, Alviandi W, Branantyo B, Daneswarry D. 2019. Validitas, reliabilitas dan adaptasi transkultural Dizziness Handicap Inventory dalam bahasa Indonesia. Oto Rhino Laryngologica Indonesiana. 49(2), 162-3. https://doi.org/10.32637/orli.v49i20.318.
- See also: Study protocol — https://perpustakaan.rsmoewardi.com/index.php?p=show_detail&id=1557

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-04-01): https://cdn.clinicaltrials.gov/large-docs/89/NCT07075289/Prot_SAP_ICF_000.pdf